CLINICAL TRIAL: NCT03032510
Title: A Phase 3, Randomized, Double-Blind, Double-Dummy, Multicenter, Prospective Study to Assess the Efficacy and Safety of IV Eravacycline Compared With Ertapenem in Complicated Urinary Tract Infections
Brief Title: Efficacy and Safety Study of Eravacycline Compared With Ertapenem in Participants With Complicated Urinary Tract Infections
Acronym: IGNITE3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tetraphase Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Organization: La Jolla Pharmaceutical Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TP-434-021
Record Dates: First submitted 2017-01-17; First posted 2017-01-26 (Estimated); Results first posted 2019-10-02 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2021-12

CONDITIONS: Complicated Urinary Tract Infections
MeSH Terms: interventions — eravacycline; Ertapenem; Levofloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Eravacycline (Intravenous)/Levofloxacin (Oral) (Experimental)
  Interventions: Drug: Eravacycline; Drug: Placebo; Drug: Levofloxacin
- Ertapenem (Intravenous)/Levofloxacin (Oral) (Active Comparator)
  Interventions: Drug: Ertapenem; Drug: Placebo; Drug: Levofloxacin

INTERVENTIONS:
Drug: Eravacycline
  Other Names: TP-434
  Arms: Eravacycline (Intravenous)/Levofloxacin (Oral)
Drug: Ertapenem
  Other Names: Invanz
  Arms: Ertapenem (Intravenous)/Levofloxacin (Oral)
Drug: Placebo
Drug: Levofloxacin
  Other Names: Levaquin

SUMMARY:
The purpose of this study is to assess the efficacy, safety, and pharmacokinetics of eravacycline compared to ertapenem in treating participants with complicated urinary tract infections (cUTI).

DETAILED DESCRIPTION:
The purpose of this study is to assess the efficacy, safety, and pharmacokinetics of eravacycline compared to ertapenem in treating participants with complicated urinary tract infections (cUTI).

This is a phase 3, randomized, double-blind, double-dummy, multicenter, prospective study to assess the efficacy, safety and pharmacokinetics of eravacycline compared with ertapenem in the treatment of cUTI.

Randomization will be stratified based on two criteria: (1) by primary site of infection (pyelonephritis and normal urinary tract anatomy vs all other diagnoses) and (2) by the receipt of a single dose of effective non-study antibiotics for the acute cUTI within 72 hours prior to randomization. An enrollment cap of approximately 50% is planned for subjects with pyelonephritis with normal urinary tract anatomy. Also, an enrollment cap of approximately 20% is planned for subjects who have received a single dose of non-study antibiotics for the acute cUTI within 72 hours prior to randomization.

In this study subjects will be enrolled and randomized to one of two treatment arms in a 1:1 ratio: (i) eravacycline intravenously (IV) / levofloxacin (PO), or (ii) ertapenem (IV) / levofloxacin (PO).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participant with either:

   1. Pyelonephritis and normal urinary tract anatomy (approximately 50% of the total population), or
   2. cUTI with at least one of the following conditions associated with a risk for developing cUTI:

      * Indwelling urinary catheter
      * Urinary retention (at least approximately 100 milliliters (mL) of residual urine after voiding)
      * History of neurogenic bladder
      * Partial obstructive uropathy (for example, nephrolithiasis, bladder stones, and ureteral strictures)
      * Azotemia of renal origin (not congestive heart failure [CHF] or volume related) such that the serum blood urea nitrogen [BUN] is elevated (>20 milligrams [mg]/deciliters [dL]) and the serum BUN:creatinine ratio is <15
      * Surgically modified or abnormal urinary tract anatomy (for example, bladder diverticula, redundant urine collection system) except urinary tract surgery within the last 30 days (placing of stents or catheters is not considered to be surgical modification)
2. At least 18 years of age at time of consent
3. Able to provide informed consent
4. At least two of the following signs or symptoms:

   1. Chills, rigors, or warmth associated with fever or hypothermia
   2. Flank pain (pyelonephritis) or pelvic pain (cUTI)
   3. Nausea or vomiting
   4. Dysuria, urinary frequency, or urinary urgency
   5. Costo-vertebral angle tenderness on physical examination
5. Urine specimen with evidence of pyuria

   1. Dipstick analysis positive for leukocyte esterase (where positive result is at least "++" as indicated on the urine dipstick provided in the laboratory kit), or
   2. ≥10 white blood cells (WBCs) per cubic millimeter, or
   3. ≥10 WBCs per high power field
6. If male: must agree to use an effective barrier method of contraception (for example, condom) during the study and for 14 days following the last dose if sexually active with a female of childbearing potential
7. If female, not pregnant or nursing or, if of childbearing potential: must commit to either use at least two medically accepted, effective methods of birth control (for example, condom, spermicidal gel, oral contraceptive, indwelling intrauterine device, hormonal implant /patch, injections, approved cervical ring) during study drug dosing and for 14 days following last study drug dose or practicing sexual abstinence

Exclusion Criteria:

1. Use of systemic antibiotics effective in cUTI within 72 hours prior to enrollment except under the following circumstances:

   1. Participants with suspected acute cUTI who have received a single dose of effective non-study antibiotics for the acute cUTI
   2. Signs and symptoms of cUTI developed while on the antibiotic for another indication
2. History of an ertapenem-resistant urinary tract infection within 1 year of enrollment
3. Likely to require >10 days of antibiotic treatment to cure the acute cUTI or likely to receive ongoing antibacterial drug prophylaxis prior to the Follow Up visit (21-28 days after randomization) [for example, participants with chronic vesiculo-ureteral reflux]
4. Unlikely to survive at least through the duration of the study
5. Hypotension, systolic blood pressure ≤90 millimeters of mercury [mmHg]
6. Complicated pyelonephritis with complete obstruction or known or suspected renal or perinephric abscess, emphysematous pyelonephritis, or Any condition likely to require surgery to achieve cure (this does not include procedure to place catheters or obtain diagnosis)
7. Known or suspected urinary fungal infection
8. Uncomplicated lower urinary tract infections
9. Suspected or confirmed active prostatitis, or currently under treatment for prostatitis
10. High risk for cUTI due to Pseudomonas (for example, history of prior cUTIs due to Pseudomonas, ≥20 mg once a day prednisone or equivalent steroid, and other risk factors as perceived by the Investigator)
11. History of renal transplantation
12. Presence of an ileal loop
13. Any history of trauma to the pelvis or urinary tract occurring within 30 days of screening
14. Indwelling urinary catheters present at screening which are not expected to be removed or replaced within 72 hours of enrollment (for example, nephrostomy tubes, stents, urethral and suprapubic catheters).
15. Known concomitant human immunodeficiency virus (HIV) infection with CD4 counts below 200 within the last six months, or an acquired immune deficiency syndrome (AIDS) defining diagnosis within the last six months
16. Neutropenia (Absolute neutrophil count <1,000 polymorphonuclear leukocytes [PMNs]/microliters [µL])
17. Participation in a study with an experimental drug or device within 30 days prior to enrollment
18. Known or suspected hypersensitivity to tetracyclines, carbapenems, or β-lactams
19. History of seizures
20. Any other unstable or clinically significant concurrent medical condition (for example, immunosuppressive therapy, chemotherapy, class IV heart or lung disease, end stage renal disease, or requiring hemodialysis) that would, in the opinion of the Investigator, jeopardize the safety of a participant and/or their compliance with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1205 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Tetraphase Pharmaceuticals
Locations (69):
- United States (10):
  - Fullerton, California
  - Los Angeles, California
  - Torrance, California
  - Coral Gables, Florida
  - Doral, Florida
  - Miami, Florida
  - Columbus, Georgia
  - St Louis, Missouri
  - Las Vegas, Nevada
  - Baytown, Texas
- Austria (3):
  - Graz
  - Linz
  - Salzburg
- Bulgaria (8):
  - Pleven
  - Plovdiv
  - Razgrad
  - Rousse
  - Smyadovo
  - Sofia
  - Varna
  - Veliko Tarnovo
- Estonia (3):
  - Tallinn
  - Tartu
  - Võru
- Georgia (2):
  - K'ut'aisi
  - Tbilisi
- Hungary (8):
  - Baja
  - Budapest
  - Miskolc
  - Nagykanizsa
  - Nyíregyháza
  - Sopron
  - Szentes
  - Tatabánya
- Latvia (3):
  - Jelgava
  - Riga
  - Valmiera
- Chisinau, Moldova
- Romania (4):
  - Brasov
  - Bucharest
  - Craiova
  - Oradea
- Russia (8):
  - Arkhangelsk
  - Moscow
  - Pyatigorsk
  - Rostov-on-the-Don
  - Saint Petersburg
  - Smolensk
  - Vsevolozhsk
  - Yaroslavl
- Slovakia (5):
  - Nitra
  - Poprad
  - Prešov
  - Svidník
  - Žilina
- Ukraine (14):
  - Chernihiv
  - Chernivtsi
  - Dnipro
  - Ivano-Frankivsk
  - Kharkiv
  - Kyiv
  - Lviv
  - Mykolaiv
  - Odesa
  - Poltava
  - Uzhhorod
  - Vinnytsia
  - Zaporizhia
  - Zhytomyr

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Eravacycline (Intravenous)/Levofloxacin (Oral): Eravacycline 1.5mg/kg IV q24h
  Placebo IV q24h
  Levofloxacin (PO)
- Ertapenem (Intravenous)/Levofloxacin (Oral): Ertapenem 1g IV q24h
  Placebo IV q24h
  Levofloxacin (PO)
Period: Overall Study
Arm/Group | Eravacycline (Intravenous)/Levofloxacin (Oral) | Ertapenem (Intravenous)/Levofloxacin (Oral)
Started | 603 | 602
Completed | 576 | 584
Not Completed | 27 | 18
Not completed — Adverse Event | 5 | 2
Not completed — Lost to Follow-up | 8 | 7
Not completed — Withdrawal by Subject | 8 | 7
Not completed — Subject noncompliance | 4 | 2
Not completed — Physician Decision | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Eravacycline (Intravenous)/Levofloxacin (Oral): Eravacycline 1.5 mg/kg IV q24h
  Placebo IV
  Levofloxacin PO
- Ertapenem (Intravenous)/Levofloxacin (Oral): Ertapenem 1.0g IV q24h
  Placebo IV
  Levofloxacin PO
- Total: Total of all reporting groups
Arm/Group | Eravacycline (Intravenous)/Levofloxacin (Oral) | Ertapenem (Intravenous)/Levofloxacin (Oral) | Total
Number analyzed (Participants) | 603 | 602 | 1205
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 338 | 331 | 669
  >=65 years | 265 | 271 | 536
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.1 (18.16) | 56.5 (19.34) | 56.8 (18.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 330 | 343 | 673
  Male | 273 | 259 | 532
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 15 | 26
  Not Hispanic or Latino | 592 | 587 | 1179
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 600 | 601 | 1201
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Latvia | 36 | 39 | 75
  Austria | 0 | 1 | 1
  Romania | 54 | 59 | 113
  Hungary | 56 | 66 | 122
  United States | 9 | 13 | 22
  Ukraine | 148 | 137 | 285
  Georgia | 33 | 40 | 73
  Slovakia | 18 | 13 | 31
  Bulgaria | 61 | 42 | 103
  Estonia | 21 | 20 | 41
  Russia | 126 | 143 | 269
  Poland | 23 | 17 | 40
  Moldova | 18 | 12 | 30

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants in the Micro-ITT Population Demonstrating Clinical Cure and Microbiologic Success at the EOI Visit
Description: This was the co-primary outcome measure for the Food and Drug Administration (FDA). The primary objective was to demonstrate the non-inferiority (NI) of eravacycline to ertapenem in responder outcome, which was derived from both clinical and microbiological responses, in the micro-ITT population. Clinical responses were either cure, failure, or indeterminate/missing; microbiological responses were characterized programmatically as either success, failure, or indeterminate/missing. Clinical cure was defined as complete resolution or significant improvement of signs or symptoms of the infection; microbiological success was a reduction of the baseline pathogen(s) to <10^4 colony-forming units/milliliter (CFU/mL). An outcome of Responder required a clinical response of cure and a microbiological response of success. Any other combination of the clinical and microbiological responses was considered either Non-responder or Indeterminate.
Time Frame: End of Infusion
Population: micro-ITT included all participants in the ITT population who had at least 1 baseline bacterial pathogen from a urine or blood culture that caused a urinary tract infection (UTI) against which eravacycline and ertapenem had expected antibacterial activity.
Measure: Count of Participants; unit: Participants
Groups:
- Eravacycline (Intravenous): Eravacycline was administered IV at a dose of 1.5 mg/kg of body weight q24h. At minimum, the first 5 doses were administered IV. An IV-to-PO transition could occur after dose 5. During PO administration, subjects received 750 mg of levofloxacin once daily. Total treatment duration was 7 or 10 days.
- Ertapenem (Intravenous): Ertapenem was administered IV at a dose of 1 g q24h. At minimum, the first 5 doses were administered IV. An IV-to-PO transition could occur after dose 5. During PO administration, subjects received 750 mg of levofloxacin once daily. Total treatment duration was 7 or 10 days.
Arm/Group | Eravacycline (Intravenous) | Ertapenem (Intravenous)
Number analyzed (Participants) | 428 | 403
Participants
  Responder | 363 | 382
  Non-responder | 51 | 7
  Indeterminate | 14 | 14

2. Primary Outcome: Proportion of Participants in the Micro-ITT Population Demonstrating Clinical Cure and Microbiologic Success at the Test-Of-Cure (TOC) Visit
Description: as for outcome 1
Time Frame: TOC visit (14-17 days after randomization)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Eravacycline; Ertapenem: micro-ITT included all participants in the ITT population who had at least 1 baseline bacterial pathogen from a urine or blood culture that caused a urinary tract infection (UTI) against which eravacycline and ertapenem had expected antibacterial activity.
Arm/Group | Eravacycline | Ertapenem
Number analyzed (Participants) | 428 | 403
Participants
  Responder | 293 | 302
  Non-responder | 116 | 86
  Indeterminate | 19 | 15

3. Secondary Outcome: Proportion of Participants in the ITT Population With Favorable Clinical Outcomes at TOC Visit
Description: Clinical cure: A complete resolution or significant improvement of signs or symptoms of the infection such that no rescue/non-study antibacterial medication was required to treat the cUTI that presented at study entry.
  Clinical failure: Subjects were classified as clinical failure in the event of
  * Death related to cUTI at any timepoint
  * Persistence of clinical symptoms of cUTI or new symptoms developed
  * Initiation of rescue/non-study antibacterial medication for cUTI Indeterminate: Study data were listed as indeterminate if the outcome was other than clinical cure or clinical failure. The reason for an indeterminate designation had to be provided Missing: Study data were listed as missing if the Investigator did not complete an assessment or if the subject did not complete the study visit.
Time Frame: TOC visit (14-17 days after randomization)
Population: ITT included all randomized participants, regardless of receiving study drug or not.
Measure: Count of Participants; unit: Participants
Groups:
- Eravacycline (Intravenous)/Levofloxacin (Oral); Ertapenem (Intravenous)/Levofloxacin (Oral): ITT included all randomized participants, regardless of receiving study drug or not.
Arm/Group | Eravacycline (Intravenous)/Levofloxacin (Oral) | Ertapenem (Intravenous)/Levofloxacin (Oral)
Number analyzed (Participants) | 603 | 602
Participants
  Clinical Cure | 547 | 566
  Clinical Failure | 31 | 20
  Indeterminate/missing | 25 | 16

ADVERSE EVENTS:
Time Frame: The time frame for adverse event reporting was from the first dose of study drug through 30 days after the last dose of study drug or the FU visit (whichever was later).
Description: The safety population was all randomized subjects who receive any amount of study drug. All safety analyses were conducted in this population and are presented by treatment actually received (not as randomized). One subject randomized to the ertapenem group received a dose of eravacycline and was included in the eravacycline group in the safety analysis.
Groups:
- Eravacycline (Intravenous): Eravacycline 1.5 mg/kg IV -The safety population was all randomized subjects who receive any amount of study drug. All safety analyses were conducted in this population and are presented by treatment actually received (not as randomized). One subject randomized to the ertapenem group received a dose of eravacycline and was included in the eravacycline group in the safety analysis.
- Ertapenem (Intravenous): Ertapenem 1 g IV-The safety population was all randomized subjects who receive any amount of study drug. All safety analyses were conducted in this population and are presented by treatment actually received (not as randomized). One subject randomized to the ertapenem group received a dose of eravacycline and was included in the eravacycline group in the safety analysis.
Arm/Group | Eravacycline (Intravenous) | Ertapenem (Intravenous)
All-Cause Mortality (participants affected / at risk) | 3/601 | 2/600
Serious Adverse Events (participants affected / at risk) | 11/601 | 6/600
Other Adverse Events (participants affected / at risk) | 174/601 | 52/600
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eravacycline (Intravenous) (N=601) | Ertapenem (Intravenous) (N=600)
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Cardiorenal syndrome (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Renal abscess (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 2 | 0
Renal colic (Renal and urinary disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Aneurysm ruptured (Vascular disorders) | 2 | 1
Circulatory collapse (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eravacycline (Intravenous) (N=601) | Ertapenem (Intravenous) (N=600)
Nausea (Gastrointestinal disorders) | 84 | 10
Vomiting (Gastrointestinal disorders) | 31 | 4
Infusion site phlebitis (General disorders) | 24 | 3
Diarrhoea (Gastrointestinal disorders) | 18 | 17
Headache (General disorders) | 17 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-07-27): https://cdn.clinicaltrials.gov/large-docs/10/NCT03032510/Prot_001.pdf
  • Statistical Analysis Plan (2018-01-22): https://cdn.clinicaltrials.gov/large-docs/10/NCT03032510/SAP_000.pdf